CLINICAL TRIAL: NCT03630783
Title: Combined Cognitive Bias Modification for Social Anxiety: A Randomized Controlled Trial
Brief Title: Combined CBM For Social Anxiety in Turkey
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Sabahattin Zaim University (Other)
Collaborators: Hacettepe University (Other)
Responsible Party: Principal Investigator, Volkan Koç, Assistant Professor, Istanbul Sabahattin Zaim University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: IstanbulSZU
Record Dates: First submitted 2018-08-02; First posted 2018-08-15 (Actual); Last update posted 2018-08-20 (Actual); Status verified 2018-08

CONDITIONS: Phobia, Social
MeSH Terms: conditions — Phobia, Social

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive Bias Modification (Group-E) (Experimental): Participants were subjected to Combined Cognitive Bias Modification in each session. During the attentional bias modification phase, photographs of neutral or threatening (disgusted) faces were used. In each trial, a pair was shown for 500 ms. Then, a sign of arrow appeared and participants were asked to indicate the direction of the arrow. In %80 of the trials, the arrow was in the same area with the neutral photograph. During the interpretational bias modification phase a threatening or positive word, as the interpretation of a sentence, appeared, then, a relevant sentence with ambiguous meaning appeared, and later, participants were asked to indicate if the word and the sentence were related. After their response a feedback (right/wrong) was given and the next trial was started.
  Interventions: Behavioral: Combined Cognitive Bias Modification
- Placebo Control (Group-C) (Placebo Comparator): Participants in this group were subjected to the same procedure as the experimental group. However, during the Combined Cognitive Bias Modification process, the sign of arrow appeared at even rates (%50 - %50) after neutral and disgusted facial impressions; and during the interpretational bias modification, sentences and relevant words were superficially related or were not related at all.
  Interventions: Behavioral: Combined Cognitive Bias Modification

INTERVENTIONS:
Behavioral: Combined Cognitive Bias Modification

SUMMARY:
In this study, it was examined whether or not combined attentional and interpretational bias modifications with university students who display social anxiety symptoms may lead to a decrease in social anxiety-related complaints. The study was conducted with 84 participants who were university students displaying social anxiety symptoms. The participants were randomly assigned into two conditions; cognitive bias modification group (E) and placebo-control group (C). Participants in group-E were subjected to attentional and interpretational bias modifications twice a week, eight sessions in total. Participants in group-C were subjected to a similar process, but without any modification. The levels of social anxiety, anxiety, depression, nonfunctional thinking of the participants were evaluated three times; just before the first session, just after the last session and two months after the last session. In addition, levels of attentional and interpretational bias of the participants were evaluated twice, just before the first session and just after the last session.

DETAILED DESCRIPTION:
A 2 (group: experimental, control) × 3 (time: pretest, posttest, follow-up) experimental design was employed. All participants were presented with informed consent form beforehand, and also verbally informed about the procedure. They were assigned to experimental (E) or attention placebo control (C) groups for 2 sessions per week, 8 sessions in total. Before the first session (pretest) and after the last session (posttest), participants were asked to answer self-report questionnaires, and their attentional and interpretational biases were assessed. And finally, participants were asked only to answer to the same questionnaires for the follow up measurements after two months.

Chi square test and independent t-test for dependent variables were run beforehand to check if participants were equally distributed to Bias Modification group-E and group-C. No statistically significant difference between group-E and group-C was observed with regards to gender distribution, social anxiety, anxiety, depression, dysfunctional thoughts, automatic thoughts, and attentional and interpretational biases.

To see the effect of 8 sessions of manipulation on attentional and interpretational bias (independent variable) created a significant difference between experimental and control groups, 2 (group: experimental [E] and control [C]) × 3 (time: pre [t1] / post [t2] / follow-up [t3]) mixed ANOVA was conducted for each dependent variable in self-report measurements, and 2 (group: experimental [E] and control [C]) × 2 (time: pre [t1] / post [t2]) mixed ANOVA were conducted for attentional and interpretational biases.

ELIGIBILITY:
Inclusion Criteria:

* Scoring above 68 on the Liebowitz Social Anxiety Scale

Exclusion Criteria:

* Having any psychiatric disorder
* Receiving a psychiatric/psychological treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2016-04 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Social anxiety | Day 0, pre-intervention
  Social anxiety symptoms were assessed with the Turkish version of the Liebowitz Social Anxiety Scale. The scale constitutes of 48 items. The lowest possible score is 48 and highest score is 192. Higher scores indicate a worse outcome.
Social anxiety | 4 weeks
  Social anxiety symptoms were assessed with the Turkish version of the Liebowitz Social Anxiety Scale. The scale constitutes of 48 items. The lowest possible score is 48 and highest score is 192. Higher scores indicate a worse outcome.
Social anxiety | 12 weeks
  Social anxiety symptoms were assessed with the Turkish version of the Liebowitz Social Anxiety Scale. The scale constitutes of 48 items. The lowest possible score is 48 and highest score is 192. Higher scores indicate a worse outcome.

SECONDARY OUTCOMES:
Depression | Day 0, pre-intervention
  Depression symptoms were assessed with the Turkish version of the Beck Depression Inventory. The scale constitutes of 21 items. The lowest possible score is 0 and highest score is 63. Higher scores indicate a worse outcome.
Depression | 4 weeks
  Depression symptoms were assessed with the Turkish version of the Beck Depression Inventory. The scale constitutes of 21 items. The lowest possible score is 0 and highest score is 63. Higher scores indicate a worse outcome.
Depression | 12 weeks
  Depression symptoms were assessed with the Turkish version of the Beck Depression Inventory. The scale constitutes of 21 items. The lowest possible score is 0 and highest score is 63. Higher scores indicate a worse outcome.
Anxiety | Day 0, pre-intervention
  Anxiety symptoms were assessed with the Turkish version of the Beck Anxiety Inventory. The scale constitutes of 21 items. The lowest possible score is 0 and highest score is 63. Higher scores indicate a worse outcome.
Anxiety | 4 weeks
  Anxiety symptoms were assessed with the Turkish version of the Beck Anxiety Inventory. The scale constitutes of 21 items. The lowest possible score is 0 and highest score is 63. Higher scores indicate a worse outcome.
Anxiety | 12 weeks
  Anxiety symptoms were assessed with the Turkish version of the Beck Anxiety Inventory. The scale constitutes of 21 items. The lowest possible score is 0 and highest score is 63. Higher scores indicate a worse outcome.
Automatic Thoughts Questionnaire | Day 0, pre-intervention
  Automatic thoughts were assessed with the Turkish version of the Automatic Thoughts Questionnaire. The scale constitutes of 30 items. The lowest possible score is 30 and highest score is 150. Higher scores indicate a worse outcome.
Automatic Thoughts Questionnaire | 4 weeks
  Automatic thoughts were assessed with the Turkish version of the Automatic Thoughts Questionnaire. The scale constitutes of 30 items. The lowest possible score is 30 and highest score is 150. Higher scores indicate a worse outcome.
Automatic Thoughts Questionnaire | 12 weeks
  Automatic thoughts were assessed with the Turkish version of the Automatic Thoughts Questionnaire. The scale constitutes of 30 items. The lowest possible score is 30 and highest score is 150. Higher scores indicate a worse outcome.
Dysfunctional Attitudes | Day 0, pre-intervention
  Dysfunctional beliefs were assessed with the Turkish version of the Dysfunctional Attitude Scale. The scale constitutes of 40 items. The lowest possible score is 40 and highest score is 280. Higher scores indicate a worse outcome.
Dysfunctional Attitudes | 4 weeks
  Dysfunctional beliefs were assessed with the Turkish version of the Dysfunctional Attitude Scale. The scale constitutes of 40 items. The lowest possible score is 40 and highest score is 280. Higher scores indicate a worse outcome.
Dysfunctional Attitudes | 12 weeks
  Dysfunctional beliefs were assessed with the Turkish version of the Dysfunctional Attitude Scale. The scale constitutes of 40 items. The lowest possible score is 40 and highest score is 280. Higher scores indicate a worse outcome.
Attentional bias | Day 0, pre-intervention
  Attentional bias was assessed with the Posner paradigm
Attentional bias | 4 weeks
  Attentional bias was assessed with the Posner paradigm
Interpretational bias | Day 0, pre-intervention
  Interpretational bias was assessed with the Word Sentence Association Paradigm
Interpretational bias | 4 weeks
  Interpretational bias was assessed with the Word Sentence Association Paradigm

CONTACTS AND LOCATIONS:
Overall Officials: Volkan Koç, PhD, Study Chair — Istanbul Sabahattin Zaim University
Locations (1):
- Volkan Koç, Küçükçekmece, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided